CLINICAL TRIAL: NCT05989490
Title: The Effect of Stretching Intensity on Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other); Research Unit for General Practice in Aalborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Intensity vs. Hypoalgesia
Record Dates: First submitted 2023-07-02; First posted 2023-08-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Pain Threshold; Stretching; Pain Sensitivity; Range of Motion
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This was a randomized, repeated-measures cross-over study. The interventions consist of two different stretching protocols (e.g., stretching to the point of discomfort and stretching to the point of pain). Subjects were randomized to one of two groups (pain first or discomfort first). Both groups underwent a static stretch protocol consisting of four bouts of thirty-second constant-angle static stretching of the knee flexors with a 20-second rest period between bouts. Subjects were instructed to keep the limb relaxed as the lower leg was passively moved towards extension to the point of discomfort and the point of pain.
Who Masked: Participant, Investigator
Masking Description: Participants were blinded to the results of all measurements and naïve to research hypotheses.
  The investigator was blinded to the results of all measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static stretching to the point of pain (Experimental): The participants are assigned to four bouts of static stretching of the right knee flexors with a 20-second rest period between bouts 20 to the point of pain.
  Interventions: Other: Static stretching
- Static stretching to the point of discomfort (Experimental): The participants are assigned to four bouts of static stretching of the right knee flexors with a 20-second rest period between bouts 20 to the point of discomfort.
  Interventions: Other: Static stretching

INTERVENTIONS:
Other: Static stretching — The participants are assigned to four bouts of static stretching of the right knee flexors with a 20-second rest period between bouts 20 to the point of discomfort and to the point of pain.

SUMMARY:
The primary objective of this study is to determine the immediate efficiency of stretching intensity on regional and distant pain sensitivity in healthy subjects. It is hypothesized that the analgesic effect of stretching may be linked with the intensity of stretching in a dose-response relationship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-55 years are recruited. As part of the screening, volunteers will also be asked to indicate known medical issues or diseases.

Exclusion Criteria:

* Participants are included if they have no known medical conditions such as; cognitive impairments, neurological, orthopaedic, or neuromuscular problems that might affect the somatosensory system or preclude stretching exercises or range of motion testing at the knee.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds | Pressure pain thresholds were measured as a baseline just prior to the induction of stretching to the point of pain and stretching to the point of discomfort
  Pressure pain thresholds was measures using a handheld pressure algometer
Pressure pain thresholds | Pressure pain thresholds were measured immediately after stretching
  Pressure pain thresholds was measures using a handheld pressure algometer

SECONDARY OUTCOMES:
Knee extension range of motion | Passive knee extension range of motion was measured as a baseline just prior to the induction of stretching to the point of pain and stretching to the point of discomfort
  Passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynamometer
Knee extension range of motion | Passive knee extension range of motion was measured immediately after stretching
  Passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynamometer
Passive resistive torque | Passive resistive torque was measured as a baseline just prior to the induction of stretching to the point of pain and stretching to the point of discomfort
  Passive resistive torque was measured using the Biodex system 4 pro isokinetic dynamometer
Passive resistive torque | Passive resistive torque was measured immediately after stretching
  Passive resistive torque was measured using the Biodex system 4 pro isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Morten P Støve, Pt. Msc, Principal Investigator — University College of Northern Denmark and Center for General Practice, Aalborg University
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data is made available upon request.
Access Criteria: Access is granted on reasonable request